CLINICAL TRIAL: NCT06379295
Title: Coronary Artery Calcification Assessed on PET Scanner (PET : Positron Emission Tomography)
Acronym: CALCOTEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHUO-2024-05
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Coronary Artery Calcification
Keywords: Coronary Disease; Coronary Artery Calcium; Cardiovascular Diseases; 18F-FDG PET/CT (Flourine-18 fluorodeoxyglucose positron emission tomography/computed tomography); Enhanced CT (computed tomography)
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Self-administered questionnaire to assess the participants risk factors, history of heart disease and medications.

SUMMARY:
Calcification artery calcium (CAC) scoring is a valuable tool for determining the risk of major adverse cardiac events.

It was found that CAC can be quantitatively assessed, by manual scoring or using deep-learning, on low-dose non electrocardiogram-gated, contrast-enhanced or non-enhanced computed tomography (CT-scan) performed in association of PET acquisition, with a good agreement with standard scans.

The purpose of this study is to determine the impact of a systematic coronary artery calcification evaluation in patients undergoing flourine-18 fluorodeoxyglucose positron emission tomography/computed tomography (18F-FDG PET/CT) imaging to improve primary prevention of cardiovascular diseases.

A visual calcification artery calcium assessment will be made for each patient, dividing them into four groups: none, mild, moderate or heavy calcification artery calcium. When possible, a calcification artery calcium score will be computed.

Each patient will complete a questionnaire to collect risk factors, history of cardiovascular diseases and medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a 18F-FDG PT/CT imaging
* Patients aged 18 and older

Exclusion Criteria:

* Patients who already participated in this study (in case of follow-up PET/CT scans)
* Unusable CT scan due to CT artifacts or poor-quality images
* Patients referred for a brain 18F-FDG PET/CT imaging
* Minors,
* Protected adults
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People aged 18 and over referred for a 18F-FDG PET/CT imaging
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of moderate calcification artery calcium (CAC) in participants without history of cardiac disease | Baseline
  In participants who had neither history of cardiac disease nor cardiology follow-up, the proportion of those with at least moderate CAC

SECONDARY OUTCOMES:
Prevalence of coronary heart disease among participants | Baseline
  Proportion of participants with history of coronary heart disease, according to questionnaire data
Correlation of CAC with the medical indication for PET imaging | Baseline
  Dividing participants into subgroups according to PET indication, determine in which subgroup the proportion of participants with at least moderate CAC is the highest
Prevalence of CAC in young participants (< 45 years old) | Baseline
  Proportion of young participants with at least mild CAC
Prevalence of moderate CAC in participants not taking low-cholesterol drug | Baseline
  In participants not taking low-cholesterol drug, proportion of them with at least moderate CAC
Prevalence of no CAC in participants taking statins | Baseline
  In participants taking statins, proportion of them without CAC

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Orléans, Orléans, France

REFERENCES:
- [Background] Agatston AS, Janowitz WR, Hildner FJ, Zusmer NR, Viamonte M Jr, Detrano R. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol. 1990 Mar 15;15(4):827-32. doi: 10.1016/0735-1097(90)90282-t. PMID 2407762
- [Background] Darby S, McGale P, Peto R, Granath F, Hall P, Ekbom A. Mortality from cardiovascular disease more than 10 years after radiotherapy for breast cancer: nationwide cohort study of 90 000 Swedish women. BMJ. 2003 Feb 1;326(7383):256-7. doi: 10.1136/bmj.326.7383.256. No abstract available. PMID 12560277
- [Background] Yeboah J, McClelland RL, Polonsky TS, Burke GL, Sibley CT, O'Leary D, Carr JJ, Goff DC, Greenland P, Herrington DM. Comparison of novel risk markers for improvement in cardiovascular risk assessment in intermediate-risk individuals. JAMA. 2012 Aug 22;308(8):788-95. doi: 10.1001/jama.2012.9624. PMID 22910756
- [Background] Hecht H, Blaha MJ, Berman DS, Nasir K, Budoff M, Leipsic J, Blankstein R, Narula J, Rumberger J, Shaw LJ. Clinical indications for coronary artery calcium scoring in asymptomatic patients: Expert consensus statement from the Society of Cardiovascular Computed Tomography. J Cardiovasc Comput Tomogr. 2017 Mar-Apr;11(2):157-168. doi: 10.1016/j.jcct.2017.02.010. Epub 2017 Feb 24. PMID 28283309
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Oh HS, Kim TH, Kim JW, Yang J, Lee HS, Lee JH, Park CH. Feasibility and limitations of deep learning-based coronary calcium scoring in PET-CT: a comparison with coronary calcium score CT. Eur Radiol. 2024 Jun;34(6):4077-4088. doi: 10.1007/s00330-023-10390-z. Epub 2023 Nov 14. PMID 37962596
- [Background] Mortensen MB, Dzaye O, Bodtker H, Steffensen FH, Botker HE, Jensen JM, Ronnow Sand NP, Maeng M, Warnakula Olesen KK, Sorensen HT, Kanstrup H, Blankstein R, Blaha MJ, Norgaard BL. Interplay of Risk Factors and Coronary Artery Calcium for CHD Risk in Young Patients. JACC Cardiovasc Imaging. 2021 Dec;14(12):2387-2396. doi: 10.1016/j.jcmg.2021.05.003. Epub 2021 Jun 16. PMID 34147446
- [Background] Pieszko K, Shanbhag A, Killekar A, Miller RJH, Lemley M, Otaki Y, Singh A, Kwiecinski J, Gransar H, Van Kriekinge SD, Kavanagh PB, Miller EJ, Bateman T, Liang JX, Berman DS, Dey D, Slomka PJ. Deep Learning of Coronary Calcium Scores From PET/CT Attenuation Maps Accurately Predicts Adverse Cardiovascular Events. JACC Cardiovasc Imaging. 2023 May;16(5):675-687. doi: 10.1016/j.jcmg.2022.06.006. Epub 2022 Sep 14. PMID 36284402
- [Background] Engbers EM, Timmer JR, Mouden M, Jager PL, Knollema S, Oostdijk AH, Ottervanger JP. Visual estimation of coronary calcium on computed tomography for attenuation correction. J Cardiovasc Comput Tomogr. 2016 Jul-Aug;10(4):327-9. doi: 10.1016/j.jcct.2016.04.002. Epub 2016 Apr 11. PMID 27089854